CLINICAL TRIAL: NCT05775718
Title: Safety and Immunogenicity of Shingrix Administered to Recipients of Allogeneic Peripheral and Cord Blood Stem Cell Transplants: Effect of Timing of Vaccination After Transplantation
Brief Title: Shingrix In Recipients of Allogeneic Transplants
Acronym: Allo
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-0394.cc; NCI-2023-04097 (Other: CTRP)
Record Dates: First submitted 2023-02-28; First posted 2023-03-20 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Bone Marrow Transplant; Stem Cell Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1-<2 years post stem cell transplant (Experimental): At Visit 1 participants will be given information about the nature of HZ and its recognition and given a questionnaire for completion should they develop HZ during the study. They will also be asked to contact the study team if they develop HZ so that further evaluation of potential HZ is completed and the details of the event recorded. A swab of an active lesion or crust from a dried lesion will be obtained for VZV PCR. A participant who develops HZ will be asked to complete the questionnaire weekly for 4 weeks and then at 8 and 12 weeks. In addition, the subject will be asked about pain medications taken during the episode. Information on HZ incidence will be supplemented from the clinic medical records and the electronic medical records. Subjects will be followed for 1 year after enrollment for the occurrence of HZ and of post-herpetic neuralgia (PHN).
  Interventions: Drug: Zoster Vaccine Recombinant
- 2-<3 years post stem cell transplant (Experimental): At Visit 1 participants will be given information about the nature of HZ and its recognition and given a questionnaire for completion should they develop HZ during the study. They will also be asked to contact the study team if they develop HZ so that further evaluation of potential HZ is completed and the details of the event recorded. A swab of an active lesion or crust from a dried lesion will be obtained for VZV PCR. A participant who develops HZ will be asked to complete the questionnaire weekly for 4 weeks and then at 8 and 12 weeks. In addition, the subject will be asked about pain medications taken during the episode. Information on HZ incidence will be supplemented from the clinic medical records and the electronic medical records. Subjects will be followed for 1 year after enrollment for the occurrence of HZ and of post-herpetic neuralgia (PHN).
  Interventions: Drug: Zoster Vaccine Recombinant
- ≥ 3 years post stem cell transplant (Experimental): At Visit 1 participants will be given information about the nature of HZ and its recognition and given a questionnaire for completion should they develop HZ during the study. They will also be asked to contact the study team if they develop HZ so that further evaluation of potential HZ is completed and the details of the event recorded. A swab of an active lesion or crust from a dried lesion will be obtained for VZV PCR. A participant who develops HZ will be asked to complete the questionnaire weekly for 4 weeks and then at 8 and 12 weeks. In addition, the subject will be asked about pain medications taken during the episode. Information on HZ incidence will be supplemented from the clinic medical records and the electronic medical records. Subjects will be followed for 1 year after enrollment for the occurrence of HZ and of post-herpetic neuralgia (PHN).
  Interventions: Drug: Zoster Vaccine Recombinant

INTERVENTIONS:
Drug: Zoster Vaccine Recombinant — Injection
  Other Names: Shingrix

SUMMARY:
This research is designed to determine if the adjuvanted recombinant glycoprotein E (gE) herpes zoster (HZ) vaccine (Shingrix) has acceptable immunogenicity and safety in people who have undergone allogeneic stem cell transplant (allo-SCT). Specifically, it will determine the effect of the interval after transplantation on the immune response and if an additional dose of vaccine is needed to improve the vaccine-induced responses.

DETAILED DESCRIPTION:
This is a phase II, single center, prospective, unblinded, immunogenicity and safety study. It is anticipated that enrollment will take approximately 6 months. Duration of participation for study subjects is approximately 1 year. During this interval, participants will continue to receive clinical care from the BMT center, which will ensure retention.

Participants will be recruited at their routine clinic visits, which take place every 6 months post-transplantation, or will be recruited by phone. Participants will be consented by study personnel in coordination with the BMT health care providers and subsequently followed in Dr. Levin's Vaccine Research Clinic, where they will also receive the 3rd dose of vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Allo-SCT recipients being age 18 - 79 years at time of allo-SCT.
* Written informed consent being obtained from the subject
* Two doses of RZV, separated by 2 to 6 months, administered at least 1 year after allo-SCT.
* Enrollment at >/= 18 months after second dose of Shingrix.
* Female subjects of childbearing potential (FOCBP) enrolled in the study only if they:

  * have practiced adequate contraception for 30 days prior to vaccination with any dose of zoster vaccine and
  * have a negative pregnancy test on the day of each dose of zoster vaccine and
  * agree to continue adequate contraception during the vaccination period and for 2 months after receipt of the vaccine.
* Investigator belief that the participant will comply with the requirements of the protocol

Exclusion Criteria:

* Active Graft Versus Host Disease (aGVHD) at the time of enrollment and receipt of the third dose of RZV
* Having received ≥20 mg prednisone for more than 2 weeks (or equivalent) in the 8 weeks preceding enrollment.
* Receiving any significant immunosuppressive therapy other than for graft maintenance, in the opinion of the investigator.
* Having received a live attenuated vaccine within the last 4 weeks, or inactivated vaccine in the last 2 weeks, prior to enrollment.
* Having a history of HZ after the administration of the primary 2-dose RZV immunization regimen.
* Pregnancy or breastfeeding
* Receiving investigational drugs from 30 day before enrollment or planned during the study
* Inability of participants unable to comply with the study schedule in the opinion of the investigator

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2028-01-20 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Compare the immune response via blood draw of Cohort 1 prior to enrollment to ≥1 year post-transplant | 1 Year
  To compare gE-specific CMI immune response of Cohort 1 in allo-SCT who received 2 doses of Shingrix ≥1 years post-transplantation and 18-30 months prior to enrollment across 3 groups defined by the time of vaccination after transplantation.
Compare the immune response via blood draw of Cohort 1 prior to enrollment to ≥1 year post-transplant to immune-competent older recipients | 1 Year
  To compare gE-specific CMI immune response of Cohort 1 in allo-SCT who received 2 doses of Shingrix ≥1 years post-transplantation and 18-30 months prior to enrollment to immunologic data previously determined in prior studies of immune-competent older recipients of RZV (age ≥50 years).
Determine adverse events after a 3rd dose of Shingrix administered 18-30 months after primary immunization for Cohort 1 | 1 Year
  Document all adverse events after 3rd dose of Shingrix.
Compare gE-specific CMI via blood draw in Cohort 1 recipients at 30-60 days after the 3rd dose of Shingrix with responses before the administration of the 3rd dose | 1 Year
  To compare gE-specific CMI in Cohort 1 recipients at 30-60 days after the 3rd dose of Shingrix with responses before the administration of the 3rd dose.
Compare gE-specific CMI via blood draw in Cohort 1 recipients at 365 days after the 3rd dose of Shingrix with responses before the administration of the 3rd dose | 1 Year
  To compare gE-specific CMI in Cohort 1 recipients at 365 days after the 3rd dose of Shingrix administered 18-30 months after the primary immunization with responses before the administration of the 3rd dose.
Compare the immune response via blood draw of Cohort 2 prior to enrollment to ≥1 year post-transplant | 1 Year
  To compare gE-specific CMI immune response of Cohort 2 in allo-SCT who received 2 doses of Shingrix ≥1 years post-transplantation and 18-30 months prior to enrollment across 3 groups defined by the time of vaccination after transplantation.
Compare the immune response via blood draw of Cohort 2 prior to enrollment to ≥1 year post-transplant to immune-competent older recipients | 1 Year
  To compare gE-specific CMI immune response of Cohort 1 in allo-SCT who received 2 doses of Shingrix ≥1 years post-transplantation and 18-30 months prior to enrollment to immunologic data previously determined in prior studies of immune-competent older recipients of RZV (age ≥50 years).
Determine adverse events after a 3rd dose of Shingrix administered 18-30 months after primary immunization for Cohort 2 | 1 Year
  Document all adverse events after 3rd dose of Shingrix.
Compare gE-specific CMI via blood draw in Cohort 2 recipients at 30-60 days after the 3rd dose of Shingrix with responses before the administration of the 3rd dose | 1 Year
  To compare gE-specific CMI in Cohort 2 recipients at 30-60 days after the 3rd dose of Shingrix administered 18-30 months after the primary immunization with responses before the administration of the 3rd dose.
Compare gE-specific CMI via blood draw in Cohort 2 recipients at 365 days after the 3rd dose of Shingrix with responses before the administration of the 3rd dose | 1 Year
  To compare gE-specific CMI in Cohort 2 recipients at 365 days after the 3rd dose of Shingrix administered 18-30 months after the primary immunization with responses before the administration of the 3rd dose.
Compare the immune response via blood draw of Cohort 3 prior to enrollment to ≥1 year post-transplant | 1 Year
  To compare gE-specific CMI immune response of Cohort 3 in allo-SCT who received 2 doses of Shingrix ≥1 years post-transplantation and 18-30 months prior to enrollment across 3 groups defined by the time of vaccination after transplantation.
Compare the immune response via blood draw of Cohort 3 prior to enrollment to ≥1 year post-transplant to immune-competent older recipients | 1 Year
  To compare gE-specific CMI immune response of Cohort 3 in allo-SCT who received 2 doses of Shingrix ≥1 years post-transplantation and 18-30 months prior to enrollment to immunologic data previously determined in prior studies of immune-competent older recipients of RZV (age ≥50 years).
Determine adverse events after a 3rd dose of Shingrix administered 18-30 months after primary immunization for Cohort 3 | 1 Year
  Document all adverse events after 3rd dose of Shingrix.
Compare gE-specific CMI via blood draw in Cohort 3 recipients at 30-60 days after the 3rd dose of Shingrix with responses before the administration of the 3rd dose | 1 Year
  To compare gE-specific CMI in Cohort 3 recipients at 30-60 days after the 3rd dose of Shingrix administered 18-30 months after the primary immunization with responses before the administration of the 3rd dose.
Compare gE-specific CMI via blood draw in Cohort 3 recipients at 365 days after the 3rd dose of Shingrix with responses before the administration of the 3rd dose | 1 Year
  To compare gE-specific CMI in Cohort 3 recipients at 365 days after the 3rd dose of Shingrix administered 18-30 months after the primary immunization with responses before the administration of the 3rd dose.
Compare gE-specific CMI via blood draw at 30-60 days after a 3rd dose of Shingrix in allo-SCT with responses of immune-competent older adults at the same time point after the dose of Shingrix | 1 Year
  To compare gE-specific CMI at 30-60 days after a 3rd dose of Shingrix in allo-SCT with responses of immune-competent older adults at the same time point after the dose of Shingrix
Compare gE-specific CMI via blood draw at 365 days after a 3rd dose of Shingrix in allo-SCT with responses of immune-competent older adults at the same time points after the 2nd dose of Shingrix | 1 Year
  To compare gE-specific CMI at 365 days after a 3rd dose of Shingrix in allo-SCT with responses of immune-competent older adults at the same time points after the 2nd dose of Shingrix.

SECONDARY OUTCOMES:
Compare gE-specific antibody responses via blood draw in allo-SCT recipients 18-30 months after primary immunization with Shingrix with responses of older immune-competent adults at 1-2 months after the administration of the primary 2-dose regimen | 1 Year
  To compare gE-specific antibody responses in allo-SCT recipients 18-30 months after primary immunization with Shingrix, and 1-2 months after the 3rd dose of Shingrix with responses of older immune-competent adults at 1-2 months after the administration of the primary 2-dose regimen.
Compare gE-specific antibody responses via blood draw in allo-SCT recipients 18-30 months after primary immunization with Shingrix with responses of immune-competent adults at 1 year after the administration of the primary 2-dose regimen | 1 Year
  To compare gE-specific antibody responses in allo-SCT recipients 18-30 months after primary immunization with Shingrix, and 1-2 months and 1 year after the 3rd dose of Shingrix with responses of older immune competent adults at 1-2 months and 1 year, respectively, after administration of the primary 2-dose regimen.
Compare VZV-specific IL2 responses via blood draw in allo-SCT recipients 18-30 months after primary immunization with Shingrix with responses of older immune-competent adults at 1-2 months after administration of the primary 2-dose regimen | 1 Year
  To compare VZV-specific IL2 responses in allo-SCT recipients 18-30 months after primary immunization with Shingrix, and 1-2 months and 1 year after the 3rd dose of Shingrix with responses of older immune-competent adults at 1-2 months and 1 year, respectively, after administration of the primary 2-dose regimen.
Compare VZV-specific IL2 responses via blood draw in allo-SCT primary immunization 1-2 months after 3rd dose of Shingrix with responses of older immune-competent adults at 1-2 months after administration of primary 2-dose response. | 1 Year
  To compare VZV-specific IL2 responses in allo-SCT recipients 18-30 months after primary immunization with Shingrix, and 1-2 months and 1 year after the 3rd dose of Shingrix with responses of older immune-competent adults at 18-30 months and 1 year, respectively, after administration of the primary 2-dose regimen.
Compare VZV-specific IL2 responses via blood draw in allo-SCT recipients 1 year after the 3rd dose of Shingrix with responses of older immune-competent adults at 1 year after administration of the primary 2-dose regimen. | 1 Year
  To compare VZV-specific IL2 responses in allo-SCT recipients 18-30 months after primary immunization with Shingrix, and 1-2 months and 1 year after the 3rd dose of Shingrix with responses of older immune-competent adults at 1-2 months and 1 year, respectively, after administration of the primary 2-dose regimen.
Compare the gE-specific T cell differentiation via blood draw in allo-SCT recipients before the 3rd dose of Shingrix to imune-competent adults | 1 Year
  To compare the gE-specific T cell differentiation in allo-SCT recipients before the 3rd dose of Shingrix with the immune profiles of immune-competent older adults before primary immunization regimen.
Compare the gE-specific T cell differentiation via blood draw in allo-SCT recipients after the 3rd dose of Shingrix to immune-competent adults | 1 Year
  To compare the gE-specific T cell differentiation in allo-SCT recipients after the 3rd dose of Shingrix with the immune profiles of immune-competent older adults after the primary immunization regimen.
Compare the gE-specific trained immunity profiles via blood draw in allo-SCT recipients before the 3rd dose of Shingrix with the profile of immune-competent adults | 1 year
  To compare the gE-specific trained immunity profiles in allo-SCT recipients before the 3rd dose of Shingrix with the immune profiles of immune-competent older adults before the primary immunization regimen.
Compare the gE-specific trained immunity profiles via blood draw in allo-SCT recipients after the 3rd dose of Shingrix with the profiles of immune-competent adults | 1 year
  To compare the gE-specific trained immunity profiles in allo-SCT recipients after the 3rd dose of Shingrix with the immune profiles of immune-competent older adults after the primary immunization regimen.
Determine the incidence of HZ in allo-SCT recipients who received 3 doses of Shingrix. | 1 year
  To assess the incidence of HZ in allo-SCT recipients who received 3 doses of Shingrix post-Tx as reported by patients.
Determine the severity of HZ via blood draw and patient dairy in allo-SCT recipients who received 3 doses of Shingrix. | 1 year
  To assess the incidence and severity of HZ in allo-SCT recipients who received 3 doses of Shingrix post-Tx as reported by patients.
Determine the predictive value of TTV titer via blood draw on the immunogenicity of the 3rd dose of Shingrix in allo-SCT | 1 year
  To assess the value of TTV titer on the immunogenicity in allo-SCT recipients who received 3 doses of Shingrix post-Tx as reported by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Myron Levin, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No